CLINICAL TRIAL: NCT03389113
Title: Effects of Whole-body Vibration Exercise on Cortical Activity and Consciousness Level in Brain Injury Patients With Minimally Conscious State: Pilot Study
Brief Title: Effects of Whole-body Vibration Exercise in Brain Injury Patients With Minimally Conscious State
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-04-101-004
Record Dates: First submitted 2017-12-27; First posted 2018-01-03 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2017-12

CONDITIONS: Brain Injuries; Minimally Conscious State
MeSH Terms: conditions — Brain Injuries; Persistent Vegetative State

STUDY DESIGN:
Intervention Model Description: Eligible patients were randomly assigned to one of the two groups in a 1:1 ratio using an odd or even random numbers table. Whole body vibration group performed five sessions of whole body vibration exercise via a vibrating platform (Galileo® Advanced Plus, Novotec Medical, Pforzheim, Germany) with a magnitude of 20 Hz and an amplitude of 4 mm. The control group performed the same sessions without vibration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole body vibration group (Experimental): Whole body vibration group performed five sessions of whole body vibration exercise via a vibrating platform (Galileo® Advanced Plus, Novotec Medical, Pforzheim, Germany) with a magnitude of 20 Hz and an amplitude of 4 mm.
  Interventions: Device: Whole body vibration; Other: Exersice
- Exercise only group (Active Comparator): The control group performed the same session without vibration.
  Interventions: Other: Exersice

INTERVENTIONS:
Device: Whole body vibration — Whole body vibration exercise is a stimulus that uses vibrations generated on a machine with oscillatory movement determined by the amplitude and frequency of the vibration.
  Arms: Whole body vibration group
Other: Exersice — Exercise maintain a half-squat position (knee joint angle at 160 degrees) on the tilt table with an incline of 60 degrees.

SUMMARY:
The purpose of this study is to investigate the effect of the whole body vibration exercise on cortical activity and consciousness Level in brain injury patients with minimally conscious state.

DETAILED DESCRIPTION:
Whole body vibration exercise can provide proper somatosensory stimulation and improve muscle strength and postural control. However, there has not yet been a report on the cortical activity changes induced by whole body vibration exercise in brain injury patients with minimally conscious state.

Patients will be randomly assigned to one of the two groups. One group will go through whole body vibration with exercise and the other will only perform exercise. The primary outcome measurement of this study was cerebral cortex activity based on changes in oxygenated hemoglobin concentration using functional near-infrared spectroscopy. Behavioral assessment were performed using the coma recovery scale-revised and modified ashworth scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose consciousness level was assessed as minimally conscious state by traumatic brain injury, stroke, and hypoxic brain injury
* Patients who had more than 3 months after brain injury

Exclusion Criteria:

* Patients under 18 years of age and older patients over 80 years
* Pregnant women
* In cases of uncontrolled internal or external disease
* Patients with severe heart, musculoskeletal problems and disabilities, and those with severe neurological lesions prior to brain injury
* Acute or chronic venous thrombosis or hemorrhage
* Person wearing an implant on the spine
* People with severe osteoporosis

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-01-02 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Cerebral cortex activity | session 0 (initial visit); session 6 (at approximately 6 days); at 2 weeks (follow-up)
  Cerebral cortex activity was measured based on changes in oxygenated hemoglobin concentration using fNIRS

SECONDARY OUTCOMES:
Coma Recovery Scale-Revised | session 0 (initial visit); session 6 (at approximately 6 days); at 2 weeks (follow-up)
  assess patients with a disorder of consciousness, commonly coma
  The CRS-R consists of 23 items, grouped into 6 sub-scales:
  1. .Auditory
  2. Visual
  3. Motor
  4. Oromotor
  5. Communication
  6. Arousal The lowest score on each sub-scale represents reflexive activity; the highest represents behaviors mediated by cognitive input.
  The total score ranges between 0 (worst) and 23 (best). This measure takes a minimum of 25 minutes to complete.
Modified Ashworth scale | session 0 (initial visit); session 6 (at approximately 6 days); at 2 weeks (follow-up)
  measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity The Ashworth scale is one of the most widely used methods of measuring spasticity, due in a large part to the simplicity and reproducible method.
  0: No increase in muscle tone Grade Description
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hee Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea